CLINICAL TRIAL: NCT07096167
Title: Advancing Pediatric Cardiovascular Health Through Afterschool Care: A Preliminary Randomized Controlled Trial
Brief Title: Afterschool Rx 2.0: Prescriptions to Afterschool Care for Pediatric Cardiovascular Risk Reduction
Acronym: ARx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Lauren von Klinggraeff, Assistant Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRBNet ID 2316862; 25CDA1451733 (Other Grant/Funding Number: American Heart Association); Career Development Award (Other Grant/Funding Number: Augusta University)
Record Dates: First submitted 2025-07-02; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Risk Factor
Keywords: cardiovascular; out-of-school time; afterschool care; pediatric; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: ORBIT Phase IIb preliminary, randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB Group (Intervention in Fall) (Other): Voucher for afterschool care and enrollment assistance provided in the fall semester, no intervention is provided in the spring semester
  Interventions: Behavioral: Voucher for Afterschool Care
- BA Group (Intervention in Spring) (Other): No afterschool voucher or enrollment assistance provided in the fall semester but is provided in the spring semester
  Interventions: Behavioral: Voucher for Afterschool Care

INTERVENTIONS:
Behavioral: Voucher for Afterschool Care — Intervention includes a voucher for afterschool care and enrollment assistance

SUMMARY:
The goal of this clinical trial is to learn if "prescribing" afterschool care to children at risk for poor heart health later in life increases their physical activity and improves their heart health. 'Prescriptions' will be provided by pediatricians at participating Federally Qualified Health Centers and vouchers to existing afterschool programs (e.g., YMCA, Boys and Girls Clubs) will be provided by the research study. The main questions this study aims to answer are:

Can afterschool care providers and health care providers easily offer and keep using the voucher program?

Will families use the voucher? Do they go to afterschool care regularly, and do the families who use them represent a wide range or backgrounds?

Does going to afterschool care help children be more physical activity?

Does going to afterschool care improve heart health?

Researchers will compare two randomly assigned time periods; one semester when families get the voucher and one semester where they do not. They will look at whether use of the afterschool care voucher leads to more physical activity and improved heart health.

ELIGIBILITY:
Inclusion Criteria:

* A child must be entering 1st-4th grade when recruited (i.e., 5-11 years old)
* A child must have one or more cardiovascular risk factors as identified by a clinical care provider (i.e., obesity, hypertension, hyperglycemia, hyperlipidemia)
* Attend an elementary school patterned with a participating afterschool program
* Belong to a family at or below 250% of the federal poverty level
* The participating parent/guardian must have a phone that accepts text messages

Exclusion Criteria:

* If the child does not meet the inclusion criteria for attending the participating afterschool programs (e.g., children that require specially trained staff to safely provide care),
* If the child is pregnant
* If it is unsafe for the child to participate in any of the study measures as determined by their clinical care provider (i.e., can not safely complete a 6-min walk test or finger stick)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of families who complete the study (RE-AIM: Individual Reach) | 9 months (end of spring semester)
  Study logs will be used to determine the proportion of families who complete the study. Participants are considered to have completed the study if they do not withdraw or drop out. A successful outcome will be considered if ≥80% of families in both groups are retained in the study and families in both sequences (AB/BA) are retained in the study at equivalent rates.
Proportion of children who attend afterschool care during intervention allocation (RE-AIM: Individual Implementation) | Baseline (beginning of fall semester) to 4 months (end of fall semester) and 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Attendance records provided by afterschool care programs will be used to determine the proportion of children who attend afterschool care during intervention allocation. Success will be defined as ≥80% of children attend afterschool care during intervention assignment.
Proportion of families that express a desire to continue attending afterschool care after the study ends (RE-AIM: Potential Maintenance) | 9 months (end of spring semester)
  Qualitative interviews with families at the school year will be used to determine families' interest in continuing to utilize afterschool care. A successful outcome will be defined as ≥80% of families in both groups express a desire to continue attending afterschool care after study ends.
Portion of clinics and clinicians that participate in prescribing afterschool care (REAIM: Setting-level Adoption) | Baseline (beginning of fall semester) , 5 months (beginning of spring semester)
  Study records will be used to measure the proportion of clinics and clinicians that prescribe afterschool care to eligible children. A successful outcome will be defined as a referral rate of ≥60% eligible children.
Proportion of afterschool programs providing afterschool care to study participants (REAIM: Setting-level adoption) | Baseline (beginning of fall semester), 5 months (beginning of spring semester)
  Study records will be used to measure the proportion of afterschool programs that are able and willing to provide afterschool care to children participating in the study. A successful outcome will be defined as having at least 8 available spots across participating programs each year (i.e., able to meet recruitment goals).
The number of days and daily hours participating afterschool programs opperate (REAIM: Setting-level Implementation) | Baseline (beginning of fall semester) to 4 months (end of fall semester) , 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Study records and random unannounced direct observation will be used to measure the number of days and daily hours the afterschool programs operate. A successful outcome will be defined as the afterschool programs being open and operational on days local elementary schools are open and operational and that the participating afterschool program follows preplanned schedule on ≥80% of observation days.

SECONDARY OUTCOMES:
Average proportion of afterschool time (14:30-19:00) spent in moderate-to-vigorous physical activity during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  An AX3 Axivity placed on children's non-dominate wrist will be used to collect minutes of afterschool time (14:30-19:00) spent in moderate-to-vigorous physical activity (data processed using Hildebrand thresholds).
Average proportion of afterschool time spent sedentary during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  An AX3 Axivity placed on children's non-dominate wrist will be used to collect minutes of afterschool time (14:30-19:00) spent sedentary (data processed using Hildebrand thresholds).
Average duration of daily screen use during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Parent-reported minutes spent using a screen (e.g., phone, computer, television) collected via electronic daily diaries will be used to calculate average duration of daily screen use.
Average sleep midpoint during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Parent-reported sleep log and Ax3 Axivity on non-dominate wrist will be used to calculate the average time halfway between sleep onset and offset (hh:mm).

OTHER OUTCOMES:
Within-person change in BMI z-score during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Age-and-sex standardized calculation of body mass index for children using height measuared in cm and weight measured in kg.
Within-person change in percent fat mass during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Change in proportion of body fat (presented as a percent, initially measured in kg)
Within-person change in blood pressure percentile during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Change in age-and-sex specific blood pressure percentile (presented as a percentile, initially measured in mmHg).
Within-person change in total cholesterol during the intervention condition compared to comparison condition | Baseline (beginning of fall semester) to 4 months (end of fall semester) VS. 5 months (beginning of spring semester) to 9 months (end of spring semester)
  Change in total cholesterol measured in mmol/L
Within-person change in HbA1c across the school year | Baseline (beginning of fall semester) to 9 months (end of spring semester)
  Change in HbA1c measured in mmol/mol

IPD SHARING:
Plan to Share IPD: Yes
Study documents including study protocols, data management procedures, and deidentified individual participate data will be made available on Open Science Framework (DOI 10.17605/OSF.IO/H7VBT).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of results with no end date